CLINICAL TRIAL: NCT03740256
Title: A First in Human Phase I Trial of Binary Oncolytic Adenovirus in Combination With HER2-Specific Autologous CAR T Cells in Patients With Advanced HER2 Positive Solid Tumors
Brief Title: Binary Oncolytic Adenovirus in Combination With HER2-Specific Autologous CAR VST, Advanced HER2 Positive Solid Tumors
Acronym: VISTA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Shalini Makawita, Assistant Professor, Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-43405 VISTA
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Bladder Cancer; Head and Neck Squamous Cell Carcinoma; Cancer of the Salivary Gland; Lung Cancer; Breast Cancer; Gastric Cancer; Esophageal Cancer; Colorectal Cancer; Pancreatic Adenocarcinoma; Solid Tumor
Keywords: HER2; Human Epidermal Growth Factor Receptor 2; Bladder; Head and Neck Squamous Cell Carcinoma; Salivary Gland; Lung; Breast; Gastric; Esophageal; Colorectal; Pancreatic; Solid Tumor
MeSH Terms: conditions — Urinary Bladder Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms; Lung Neoplasms; Breast Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Phase (Experimental): Five dose levels will be evaluated using the BOIN design. Cohorts of size 3 will be enrolled at each dose level until 9 evaluable patients have been studied at a single dose. Each patient will receive an intratumoral injection of CAdVEC alone on Day 1 or combined with an injection of HER2.CAR.T cells on Day 4, according to the following dose levels:
  Dose Level 1 CAdVEC = 5.00E+9 HER2 specific CAR-T cells = 0
  Dose Level 2 CAdVEC = 1.00E+10 HER2 specific CAR-T cells = 0
  Dose Level 3 CAdVEC = 1.00E+10 HER2 specific CAR-T cells = 1.00E+06
  Dose Level 4 CAdVEC = 1.00E+10 HER2 specific CAR-T cells = 1.00E+07
  Dose Level 5 CAdVEC = 1.00E+10 HER2 specific CAR-T cells = 1.00E+08
  Interventions: Biological: CAdVEC

INTERVENTIONS:
Biological: CAdVEC — The intratumoral administration of CAdVEC will create a pro-inflammatory tumor microenvironment and will promote the recruitment and expansion of adoptively transferred HER2 specific CAR T cells via CAR (tumor antigen). We expect HER2 CAR T cells expanded at primary tumor sites will re-circulate and target metastasized tumors. The combination we propose to test has the potential to overcome each of the established individual limitations of oncolytic viruses and of CAR T-cells. Testing each element separately would not be beneficial or informative, since the combination therapy is anticipated to have unique profiles of both therapeutic benefit and potential toxicities.
  Other Names: HER2-specificCAR- T

SUMMARY:
This study is a first in human Phase 1 study that involves patients with a type of cancer called HER2 (Human Epidermal Growth Factor Receptor 2) positive cancer.

This study asks patients to volunteer to take part in a research study investigating the safety and efficacy of using special immune cells called HER2 chimeric antigen receptor specific cytotoxic T lymphocytes (HER2 specific CAR T cells), in combination with intra-tumor injection of CAdVEC, an oncolytic adenovirus that is designed to help the immune system including HER2 specific CAR T cell react to the tumor.

The study is looking at combining these two treatments together, because we think that the combination of treatments will work better than each treatment alone. We also hope to learn the best dose level of the treatments and whether or not it is safe to use them together.

In this study, CAdVEC will be injected into participants tumor at one tumor site which is most easiest to reach. Once it infects the cancer cells, activation of the immune response will occur so it can attack and kill cancer cells. (This approach may have limited effects on the other tumor sites that have not received the oncolytic virus injection, so, patients will also receive specific T cells following the intratumor CAdVEC injection.) These T cells are special infection-fighting blood cells that can kill cells infected with viruses and tumor cells.

Investigators want to see if these cells can survive in the blood and affect the tumor. Both CAdVEC and HER2-specific autologous CAR T are investigational products. They are not approved by the FDA.

DETAILED DESCRIPTION:
Treatment with CAdVEC:

On the first day of treatment, participants will receive an injection of CAdVEC into their tumor.

A blood sample will be obtained from the participant before the CAdVEC intratumor injection . Depending on the location of the tumor, different techniques can be used for the injection into your tumor. The most common route of injection is ultrasound-guided percutaneous (needle puncture in the skin) injection, but endoscopic (using a lighted, flexible instrument called an endoscope) ultrasound-guidance will be used for some patients as appropriate. Prior to percutaneous injection, participants may receive an anti-anxiety medicine to calm them down, to relieve muscle spasms, and provide sedation. If the participants tumor is injected during an endoscopic procedure, the procedure may be done under sedation.

Treatment with HER2- specific autologous T Cells:

The participant will have given blood earlier for us to make HER2 targeting cytotoxic T-lymphocytes (HER2- specific autologous T Cells). These cells are grown in the lab and frozen for participants. Investigators make the cells by combining dendritic cells (DCs) or monocytes with the T cells in the presence of produced mixtures of adenoviral proteins. Investigators then put a new gene in to those T cells to make them specifically attract to and kill HER2 positive tumors. As the T cells grow, they are cultured by adding adenoviral proteins for stimulation and expansion. Investigators call those T cells: HER2- targeting T cells (HER2- specific autologous T Cells).

This study looks at different doses of HER2- specific autologous T Cells. The decision about the dose participants receive is determined when enrolled on the study.

Five dose levels will be evaluated. Cohorts of size 3 will be enrolled at each dose level until 9 evaluable patients have been studied at a single dose. Each patient will receive an intratumoral injection of CAdVEC alone on Day 1 or combined with an injection of HER2.CAR T cells on Day 4.

CAdVEC intratumoral injection will be given as a single injection to a single appropriate tumor site by direct, endoscopic, or image-guided injection on Day 1. After receiving the CAdVEC injection participants will be observed for 2-4 hours before leaving the hospital. During that time the study team will monitor vital signs and watch for any side-effects from the treatment. Participants will also be contacted by telephone about 24 hours after receiving the CAdVEC injection.

HER2.CAR T cells will be given intravenously on day 4 after CAdVEC injection, with a 3 day window (until day 7).

Before receiving the T cell infusion, participants may be given Benadryl (diphenhydramine) and Tylenol (acetaminophen). Tylenol and Benadryl are given to prevent a possible allergic reaction to the T cell administration. After receiving the infusion of HER2-specific autologous T cells participants will be observed for at least 3 hours before they may leave the hospital. Additionally, participants must plan to remain in the Houston area for at least 3 weeks after the infusion.

Standard medical tests before treatment:

Before being treated, participants will receive a series of standard medical tests and procedures as well as research blood draws.

Standard Medical tests during and after treatment:

During treatment, participants will receive standard medical tests and procedures as well as research blood draws.

Study specific evaluations:

Investigators will follow participants closely after treatment for any side effects for at least 2 years after the last infusion.

To learn more about the way the T cells are working in the body, an extra blood sample will be taken before the CAdVEC injection, before the CAR T cell infusion, and at week 1, 2, 4 , 6, months 3, 6, 9 and 12 after CAR T cell infusion. Thereafter every 6 months up to 5 years and then yearly for 15 years. Investigators will use this blood to see how long the T cells last and to look at the immune response to the cancer. Investigators may also obtain a tumor tissue biopsy before CAdVEC injection, between days 5 and 10 after infusion of the HER-2 CAR-T cells, and at the time tumor recurs. Urine will be collected before CAdVEC injection, Days 2, 4 (or the day of CAR T-cell infusion), weeks 1 and 2 after CAR T cell infusion.

ELIGIBILITY:
Inclusion Criteria:

This study will look at solid tumors (as a basket trial for any solid cancer) with HER2 positivity based on IHC

Procurement Inclusion Criteria

1. The patient has a histologically confirmed advanced refractory HER2 positive solid tumor, including but not limited to: head and neck squamous cell carcinoma; cancer of the salivary glands; lung cancer; breast cancer; bladder cancer; gastric cancer; esophageal cancer; colorectal cancer; and pancreatic adenocarcinoma. HER2 positivity is defined as ≥2+ staining by IHC with either the FDA-approved CB11 antibody (Leica) or anti HER2/neu (4B5) (VENTANA), which refers to greater than weak-to-moderate staining intensity in >10% tumor cells.
2. The disease must be deemed unsuitable for curative treatments including surgery, radiotherapy, systemic therapy, including checkpoint inhibitors, or any combination of the above modalities by the referring oncology physician and confirmed by the senior oncologists leading the protocol.
3. Disease must have progressed after standard first line therapy, or without available effective treatment options. Patients are still eligible if they have failed more than one line of therapy.
4. The patient must have at least one tumor site appropriate for intratumoral injection.
5. The patient must have radiographically measurable disease as per RECIST 1.1.
6. Life expectancy more than 12 weeks.
7. The patient is ≥ 18 years of age, able to understand and give informed consent to study related procedures and treatments.

Procurement Exclusion Criteria

1. History or evidence of active autoimmune disease requiring continuous systemic corticosteroids (with more than 10mg/day prednisone or equivalent dose), immunosuppressants or other disease modifying agents (except palliative radiation).
2. Evidence of significant immunosuppressive conditions, such as the following:

   * Post organ transplant.
   * Diagnosis of HIV or other immunodeficiency disorders.
3. Diagnosis of other malignancies within 5 years except for cutaneous basal cell or squamous cell carcinoma, well-differentiated thyroid cancer, or localized prostate cancer.
4. Patients with known active hepatitis B or C infection.
5. Patient has had acute myocardial infarction within 6 months prior to consent for procurement.
6. Injectable tumor site is considered to incur a significant risk of major hemorrhage (e.g. located in the CNS (brain), and proximal to critical neurovascular structures) per investigator's review.
7. Uncontrolled intercurrent illness including but not limited to psychiatric illness and or social situations that in the opinion of the investigator would compromise compliance of study requirements or put the patient at unacceptable risk.

Treatment Inclusion Criteria:

1. Histologically confirmed advanced refractory HER2 positive solid tumors, including but not limited to: head and neck squamous cell carcinoma; cancer of the salivary glands; lung cancer; breast cancer; bladder cancer; gastric cancer; esophageal cancer; colorectal cancer; and pancreatic adenocarcinoma. HER2 positivity is defined as ≥2+ staining by IHC with either the FDA-approved CB11 antibody (Leica) or anti HER2/neu (4B5) (VENTANA), which refers to greater than weak-to-moderate staining intensity in >10% tumor cells (HER2 positivity requirement is excluded in DL1 and DL2 as HER2 targeted agents are not used).
2. The disease must be deemed unsuitable for curative treatments including surgery, radiotherapy, systemic therapy, including checkpoint inhibitors, or any combination of the above modalities by the referring oncology physician and confirmed by the senior oncologists leading the protocol.
3. Disease must have progressed after standard first line therapy, or without available effective treatment options. Patients are still eligible if they have failed more than one line of therapy.
4. The patient must have at least one tumor site appropriate for intratumoral injection.
5. The patient must have radiographically measurable disease as per RECIST 1.1.
6. The patient must have adequate organ function within 7 days prior to treatment as indicated by following measures:

   * Hematologic: Absolute neutrophil count (ANC) ≥1.0 x 10^9/l; Hemoglobin ≥7 g/dl; Platelet count ≥ 100 x 10^9/l; PT or PTT ≤ 1.5 x ULN unless the subject is receiving anticoagulation.
   * Hepatic function: bilirubin < 2 x ULN, and AST and ALT < 3 x ULN
   * Renal Function: serum creatinine <2 x the ULN or creatinine clearance >60 mL/min.
7. Prior HER2 targeted therapy is allowed if delivered at least 4 weeks prior to the enrollment. (Excluding DL1 and DL2)
8. Eastern Cooperative Oncology Group (ECOG) performance status 2 or less (Appendix I).
9. Females of childbearing potential must have a negative pregnancy test and agree to use contraception during on-study protocol therapy, or deemed to be not able to get pregnant.
10. Male subjects with pregnant partner/female partner of childbearing potential agree to use barrier contraceptive during the study to minimize the risk of embryo-fetal exposure.
11. The patient is ≥ 18 years of age, and able to understand and give informed consent to study related procedures and treatments.

Treatment Exclusion Criteria:

1. Patients with any concurrent treatment that would compromise the study including but not limited to continuous high dose corticosteroids (more than 10mg/day prednisone or equivalent dose), lympho-depleting antibodies, immunotherapy, targeted therapies or cytotoxic agents, CNS metastasis requiring continuous high-dose steroids (more than 10mg/day prednisone or equivalent dose) or other active therapeutic intervention. This does not include stable, previously-treated brain metastases. Patients on DL1 and DL2 can continue prior checkpoint inhibitors and HER2 targeted agents during the DLT evaluation period.
2. Patients at significant risk of airway compromise or other critical obstruction (e.g. bowel, ureter, etc.) in the event of possible post injection tumor inflammation based on the investigative team's judgement.
3. History or evidence of active autoimmune disease requiring continuous systemic corticosteroids, immunosuppressants or other disease modifying agents.
4. Evidence of significant immunosuppressive conditions, such as the following:

   * Post organ transplant.
   * Diagnosis of HIV or other immunodeficiency disorders.
5. Diagnosis of other malignancies within 5 years except for cutaneous basal cell or squamous cell carcinoma, well-differentiated thyroid cancer, or localized prostate or cervical cancer.
6. Patients with known active infectious disease, such as hepatitis B or C infection.
7. Patient has had acute myocardial infarction within 6 months prior to enrollment for treatment.
8. Patients with abnormal left ventricular function (LVEF <55%).
9. Injectable tumor site is considered to incur a significant risk of major hemorrhage (e.g. located in the CNS (brain), pulmonary parenchyma, and proximal to critical neurovascular structures).
10. Pregnant or breastfeeding females.
11. Uncontrolled intercurrent illness including but not limited to psychiatric illness and or social situations that in the opinion of the investigator would compromise compliance of study requirements or put the patient at unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2038-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity (DLT) by CTCAE 5.0 | 4 weeks after the HER2.CAR AdVST infusion or 4 weeks + 3 days after the CAdVEC injection.
  Incidence of dose limiting toxicities (DLT) of CAdVEC intratumoral injection in combination with HER2.CAR AdVST cells in patients with advanced refractory HER2 positive solid tumors.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) according to RECIST1.1 criteria | 13 weeks
  Overall response rate is defined as the number of patients experiencing PR or better (i.e. PR + CR) divided by the number evaluable for efficacy. Tumor regression or progression will be evaluated accordingly with RECIST 1.1 criteria.
Disease Control Rate (DCR) | 13 weeks
  Disease Control Rate is defined as as the number of patients experiencing SD or better (i.e. SD+PR+CR) divided by the number evaluable for efficacy. Tumor regression or progression will be evaluated accordingly with RECIST 1.1 criteria.
Progression Free Survival (PFS) | 15 years
  Progression-Free Survival is defined as the time from start of treatment to disease progression or death.
Overall Survival (OS) | 15 years
  Overall survival is defined as the time from the start of treatment to death due to any cause.
Number of treatment related adverse events with grade 3 or greater severity by CTCAE 5.0 | 30 days
  Treatment related adverse events with grade 3 or greater severity by CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Makawita, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor St. Luke's Medical Center, Houston, Texas, United States